CLINICAL TRIAL: NCT00133549
Title: Evaluation of a 9-valent CRM 197- Conjugated Pneumococcal Polysaccharide Vaccine in Elderly Adults
Brief Title: 9-valent CRM 197 Pneumococcal
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 99-023
Record Dates: First submitted 2005-08-19; First posted 2005-08-23 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2011-05

CONDITIONS: Pneumococcal Infection
Keywords: pneumococcal vaccine, 23-valent polysaccharide vaccine, elderly
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 2 (Experimental): Vaccine dose 1: CRM-PS; Vaccine dose 2 (month 4): CRM-PS; Vaccine dose 3 (month 8): PS.
  Interventions: Biological: PNU-IMUNE®23; Biological: Nine-valent pneumococcal conjugate (PNCRM9)
- 1 (Experimental): Vaccine dose 1: CRM-PS; Vaccine dose 2 (month 4): saline placebo; Vaccine dose 3 (month 8): PS.
  Interventions: Drug: Placebo; Biological: PNU-IMUNE®23; Biological: Nine-valent pneumococcal conjugate (PNCRM9)
- 3 (Active Comparator): Vaccine dose 1: PS; Vaccine dose 2 (month 4): saline placebo; Vaccine dose 3 (month 8): saline placebo.
  Interventions: Drug: Placebo; Biological: PNU-IMUNE®23

INTERVENTIONS:
Drug: Placebo — Saline placebo administered in a volume of 0.5 ml intramuscularly.
  Arms: 1; 3
Biological: PNU-IMUNE®23 — The 23-valent pneumococcal vaccine (PS) vaccine will contain a mixture of 25 micrograms purified, pneumococcal polysaccharide of each of 23 serotypes of Streptococcus pneumoniae per 0.5 ml dose in isotonic saline and 0.01% thimerosal. The vaccine will be administered in a volume of 0.5 ml intramuscularly.
Biological: Nine-valent pneumococcal conjugate (PNCRM9) — Cross-reactive material 197 (CRM 197) is a product of the Corynebacterium diphtheria C7. Vaccine is prepared from pneumococcal polysaccharides of types 1, 4, 5, 9V, 14, 18C, 19F, 23F (2 mcg each) and 6B (4 mcg) covalently linked to CRM197 by reductive amination. The protein-polysaccharide combination is prepared as a lyophilized powder with aluminum phosphage which is reconsitituted before use. The vaccine will be administered in a volume of 0.5 ml intramuscularly.
  Arms: 1; 2

SUMMARY:
The purpose of this study is to evaluate the safety and immune response of a conjugated pneumococcal vaccine compared to a licensed 23-valent polysaccharide pneumococcal vaccine in elderly adults. Study participants will include 180 adults, 65 years of age or greater. Participants will be randomly assigned to 1 of 3 possible groups. Subjects will maintain a study diary to record side effects and oral temperatures for 7 days following each vaccination. Blood samples will be collected before and 1 month following each dose of vaccine or placebo. Participants will be involved in study related procedures for up to 268 days.

DETAILED DESCRIPTION:
Elderly individuals are at an increased risk for serious pneumococcal infection. The efficacy of the licensed pneumococcal vaccine is also lower in this at risk population. The precise immunologic reason for the increased susceptibility and decreased efficacy with advancing age is unknown. Understanding and improving the response to pneumococcal vaccine in persons over the age of 65 is an important step in preventing this serious illness. The proposed study will evaluate the relative safety and immunogenicity of 9-valent CRM 197 protein-conjugated pneumococcal polysaccharide (CRM-PS) compared to the currently licensed 23-polysaccharide (PS) vaccines in elderly adults. In addition, the response to revaccination following conjugate vaccine will also be evaluated. Outcome measurements will include adverse effects, standard ELISA measurements of serotype specific antibody, as well as antibody response to carrier protein, effects on functional antibody status and on nasal carriage of S. pneumoniae. The study will be conducted in 180 adults who are 65 years of age and older and who have not received pneumococcal vaccine within the last 5 years. Patients will be assigned to 1 of 3 groups at random in a double blind manner. One dose of vaccine and 1 dose of placebo or 2 doses of 9-valent CRM-PS vaccine will be administered at an interval of 4 months and compared to a single dose of PS vaccine and 1 dose of placebo. Subjects will be evaluated for local and system side effects using a 7-day diary card and clinical and telephone follow-up. Serologic evaluation will be done before and 1 month following each vaccination or placebo. Subjects who received CRM-PS will receive a dose of PS vaccine 8 months after the first dose of vaccine, and potential priming by previous conjugate vaccine will be assessed by measuring the quality and quantity of the antibody response to revaccination. Participants will be involved in study related procedures for up to 268 days.

ELIGIBILITY:
Inclusion Criteria:

* Persons age 65 years and older.
* Able to give informed consent. Informed consent will be assessed with a brief questionnaire.
* Subjects must be physically able to monitor and record side effects, including reading a digital thermometer and measuring erythema and induration, with assistance from others as needed.
* Subjects must be available for follow-up over the next 9 months

Exclusion Criteria:

* Known previous receipt of licensed pneumococcal PS vaccination within the previous 5 years. Prior vaccination history will be obtained from current and previous health care providers, if available.
* Previous vaccination with any pneumococcal glycoconjugate vaccine.
* High risk medical condition for pneumococcus such as splenectomy, nephrotic syndrome, or lymphoma.
* Immunosuppressive diseases or immunosuppressive therapy. This includes doses of steroids greater than 10 mg daily (or its equivalent), cancer chemotherapy, or known HIV disease.
* History of idiopathic thrombocytopenic purpura.
* Acute respiratory illness or fever (temperature >38 degrees C or 100.4 degrees F) within one week of vaccination. Subjects can be reconsidered for enrollment when they recover from their illness.
* History of allergy to any of the vaccine components or previous severe allergic reaction to any vaccination.
* Any medical condition that would in the opinion of the investigator, interfere with the evaluation of the study objectives.
* Documented S. pneumoniae infection in the past 5 years.
* Screening laboratory values outside the following limits: 1) hematocrit below 28%, 2) WBC <3,000 or over 13,500 per ul, 3) platelets below 125,000 or above 500,000 per ul, 4) creatinine above 2.8 mg/dl or BUN above 75 mg/dl, and 5) AST/SGOT or ALT/SGPT over 110 U/L, Alkaline phosphatase over 200 IU/I or a bilirubin over 2.8 mg/dl.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 180 (Actual)
Dates: Start 2000-11; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Adverse effects. | Duration of study.
Antibody response to carrier protein, effects on functional antibody status and on nasal carriage of S. pneumoniae. | Before and 1 month following each vaccine or placebo.
Standard ELISA measurements of serotype specific antibody. | Before and 1 month following each vaccine or placebo.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Rochester, Rochester, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio